CLINICAL TRIAL: NCT03674762
Title: Submerged vs. Nonsubmerged Single Laser-microgrooved Implants. Clinical and Radiographic Results at 3-years of RCT With Split Mouth Design.
Brief Title: Submerged vs. Nonsubmerged Single Laser-microgrooved Dental Implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Renzo Guarnieri, professor, University of Roma La Sapienza
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4597
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Partially Edentulous Maxilla, Mandible
Keywords: submerged two-stage, nonsubmerged one-stage, dental implants, marginal bone loss

STUDY DESIGN:
Intervention Model Description: The cases were randomly divided into two groups as two-stage/submerged, and one-stage/nonsubmerged. Thus, in each patient, the two implants (submerged and nonsubmerged) were placed randomly in the left and right hemi-mandible or in the left and right hemi-maxilla
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dental implants (Experimental): microgrooved dental implants submerged
  Interventions: Device: Microgrooved dental implants
- dentale implants (Experimental): microgrooved dental implants nonsubmerged
  Interventions: Device: Microgrooved dental implants

INTERVENTIONS:
Device: Microgrooved dental implants — Dental Implant placement

SUMMARY:
Aim: to evaluate and compare radiographic marginal bone loss (MBL) and soft tissue parameters around submerged/two-stage and nonsubmerged/one-stage single implants with same tapered body design and surface, same thread design and distance, and same collar surface (laser-microgrooved), after 3 years of loading.

DETAILED DESCRIPTION:
Materials and methods: 20 submerged/two-stage implants and 20 nonsubmerged/one stage implants were placed randomly with a split mouth design, in 20 partially edentulous patients. Radiographic and clinical examinations were carried out at the implant placement (Baseline, BSL), at the delivery of prosthetic restorations (T0), and at each year of the follow-up period (T1, T2, T3). Plaque index (PI), probing depth (PD), bleeding on probing (BOP), and gingival recession (REC) were recorded. Radiographic marginal bone levels (MBL) were assessed at the mesial (MI) and distal (DI) aspect of implant sites. In addition, the influence of keratinized tissue thickness (KTT) on MBL was investigated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were: age ≥ 18 years, good general health, without contraindications to implant surgery, presence of at least two non-adjacent edentulous sites requiring implant therapy. Each implant site had to be located in the left or right hemi-posterior mandible or in the left or right hemi- posterior maxilla.

-

Exclusion Criteria:

* Exclusion criteria were: implants placed into regenerated bone, lack of a periodontal chart and periapical radiograph at the beginning and at the end of follow-up period, alcohol and drug abuse, pregnancy, or uncontrolled metabolic disorders, tobacco smoking (> 10 cigarettes/day), full mouth plaque score (FMPS), and full mouth bleeding score /FMBS) ≥25%, periodontally compromised patients (with attachment loss of 3 mm and/or radiographic bone loss of 30% of root length in 30% of sites), teeth adjacent to the implant area (mesial and distal) affected by untreated periodontal and/or endodontic infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
radiographic marginal bone loss | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universita la Sapienza, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esposito M, Coulthard P, Thomsen P, Worthington HV. Interventions for replacing missing teeth: different types of dental implants. Cochrane Database Syst Rev. 2005; 1:CD003815 Brånemark PI, Hansson BO, Adell R, Breine U, Lindström J, Hallén O, et al. (1977) Osseointegrated implants in the treatment of the edentulous jaw. Scandinavian Journal of Pasticic and Reconstructive Surgery; 16: 1-99. . Akcali A, Trullenque-Eriksson A, Sun C, Petrie A, Nibali L, & Donos N. (2017) What is the effect of soft tissue thickness on crestal bone loss around dental implants? A systematic review. Clinical Oral Implant Research; 28, 1045-1053. Becktor JP, Isaksson S, Billström C. (2007) A prospective multicenter study using two different surgical approaches in the mandible with turned Brånemark implants: Conventional loading using fixed prostheses. Clinical Implant Dentistry and Related Research ;9:179-185. Berglundh T, Abrahamsson I,Welander M, Lang NP, Lindhe J. (2007) Morphogenesis of the peri-implant mucosa: An experimental study in dogs. Clinical Oral Implant Research; 18:1-8. Broggini N, McManus LM, Hermann JS, Medina RU, Oates TW, Schenk RK, et al. (2003). Persistent acute inflammation at the implant-abutment interface. Journal of Dental Research 82:232-237. Buser D, Mericske-Stern R, Bernard JP, et al. (1997) Long-term evaluation of non-submerged ITI implants. Part 1: 8-year life table analysis of a prospective multi-center study with 2359 implants. Clinical Oral Implants Research; 8:161-172. Cecchinato D, Olsson C, Lindhe J. (2004) Submerged or non-submerged healing of endosseous implants to be used in the rehabilitation of partially dentate patients. Journal of Clinical Periodontoly ;31:299-308. Cordaro L, Torsello F, Roccuzzo M (2009). Clinical outcome of submerged vs. non-submerged implants placed in fresh extraction sockets. Clinical Oral Implants Research ;20:1307-1313. Esposito M, Coulthard P, Thomsen P, Worthington HV. (2005) Interventions for replacing missing teeth: different types of dental implants. The Cochrane Database of Systematic Reviews; 1:CD003815 Esposito M, Grusovin MG, Chew YS, Coulthard P, Worthington HV. (2009) One-stage versus two-stage implant placement. A Cochrane systematic review of randomised controlled clinical trials. European Journal of Oral Implantology. Summer;2(2):91-9. Hermann, J.S., Cochran, D.L., Nummikoski, P.V. & Buser, D. (1997) Crestal bone changes around titanium implants. A radiographic evaluation of unloaded non-submerged and submerged implants in the canine mandible. Journal of Periodontology 68: 1117-1130. Jansen, V.K., Conrads, G. & Richter, E.-J. (1997) Microbial leakage and marginal fit of the implant-abutment interface. International Journal of Oral and Maxillofacial Implants 12: 527-540 Jung RE, Jones AA, Higginbottom FL, Wilson TG, Schoolfield J, Buser D, Hämmerle CH, Cochran DL (2008) The influence of nonmatching implant and abutment diameters on radiographic crestal bone levels in dogs. Journal of Periodontology. Feb;79(2):260-70. Linkevicius T, Apse P, Grybauskas S, & Puisys A. (2009) The influence of soft tissue thickness on crestal bone changes around implants: A 1-year prospective controlled clinical trial. International Journal of Oral & Maxillofacial Implant; 24, 712-719. Linkevicius T, Apse, P, Grybauskas S, & Puisys A. (2010) Influence of thin mucosal tissues on crestal bone stability around implants with platform switching: A 1-year pilot study. Journal of Oral & Maxillofacial Surgery; 68, 2272-2277.
- [Derived] Guarnieri R, Di Nardo D, Di Giorgio G, Miccoli G, Testarelli L. Clinical and radiographics results at 3 years of RCT with split-mouth design of submerged vs. nonsubmerged single laser-microgrooved implants in posterior areas. Int J Implant Dent. 2019 Dec 18;5(1):44. doi: 10.1186/s40729-019-0196-0. PMID 31848762